CLINICAL TRIAL: NCT01938183
Title: Full-mouth Periodontal Debridement With or Without Adjunctive Metronidazole Gel in Smoking Patients With Chronic Periodontitis
Brief Title: Full-mouth Periodontal Debridement and Metronidazole Gel in Patients With Chronic Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Francisco Groppo, Full Professor, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTZ085-2006
Record Dates: First submitted 2013-08-30; First posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Periodontitis
Keywords: chronic periodontitis; metronidazole
MeSH Terms: conditions — Chronic Periodontitis | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Full-mouth PD+placebo gel (Placebo Comparator): Full-mouth periodontal debridement using an ultrasonic device in a single session for approximately 1 hour + trays with 3 g of placebo gel (semi-solid suspension containing carbopol), overnight, during seven days.
  Interventions: Procedure: Full-mouth periodontal debridement; Drug: placebo gel
- Full-mouth PD+Metronidazole tablet (Active Comparator): Full-mouth periodontal debridement using an ultrasonic device in a single session for approximately 1 hour + single oral dose of 750 mg tablets/day at night, during seven days.
  Interventions: Procedure: Full-mouth periodontal debridement; Drug: Metronidazole tablet
- Full-mouth PD+Metronidazole benzoate gel (Active Comparator): Full-mouth periodontal debridement using an ultrasonic device in a single session for approximately 1 hour + trays with 3 g of 15% Mtz benzoate gel (semi-solid suspension containing carbopol), overnight, during seven days.
  Interventions: Procedure: Full-mouth periodontal debridement; Drug: Metronidazole benzoate gel

INTERVENTIONS:
Procedure: Full-mouth periodontal debridement — full-mouth periodontal debridement using an ultrasonic device in a single session for approximately 1 hour
  Other Names: PD
Drug: Metronidazole tablet — 750 mg metronidazole tablets
  Other Names: MTZ tablet
  Arms: Full-mouth PD+Metronidazole tablet
Drug: placebo gel — semi-solid suspension containing carbopol
  Arms: Full-mouth PD+placebo gel
Drug: Metronidazole benzoate gel — 15% Mtz benzoate in semi-solid suspension containing carbopol (gel)
  Other Names: MTZ GEL
  Arms: Full-mouth PD+Metronidazole benzoate gel

SUMMARY:
Hypothesis: metronidazole gel applied topically after periodontal debridement in smokers volunteers could improve clinical parameters when compared to metronidazole tablets + periodontal debridement. Method: 30 smokers with chronic periodontitis were randomly assigned into 3 groups: periodontal debridement combined with 3 g placebo gel; periodontal debridement combined with daily topical application of 3 g metronidazole benzoate gel (15%); and periodontal debridement combined with a daily single dose of 750 mg metronidazole. Clinical parameters evaluated were visible plaque, gingival bleeding, probing pocket depth and relative attachment level.

DETAILED DESCRIPTION:
Background. The benefit of adjunctive metronidazole on periodontal procedure in smokers with chronic periodontitis (CP) is uncertain. The authors compared the effect of metronidazole (Mtz) on full-mouth periodontal debridement (PD= 1 hour of ultrasonic calculus/plaque removal) in smokers with CP.

Methods. This pilot study involved 30 Individuals (having at least six teeth with a clinical attachment loss of ≥ 5 mm and probing pocket depth (PPD) of ≥5 mm) that were randomly assigned into three groups (n=10): 1) PD plus 3 g of placebo gel daily topical application 2) PD plus daily topical application of 3 g of 15% Mtz benzoate gel; and 3) PD plus a daily single dose of 750 mg Mtz (Flagyl®). Clinical parameters visible plaque index (VPI), gingival bleeding index (GBI), relative attachment level (RAL) and PPD; and the quantitative analysis (real-time PCR) of Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis and Tannerella forsythia were assessed baseline, 1, 3 and 6 months after PD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic periodontitis
* presence of at least 6 periodontal pockets with a clinical attachment loss of ≥5 mm
* bleeding on probing (BOP)
* radiographic bone loss
* probing pocket depth higher or equal to 5 mm in at least six teeth
* at least 20 teeth in mouth (third molars excluded)
* an established smoking habit (at least 10 cigarettes per day for the past 4 years)

Exclusion Criteria:

* periapical alterations in qualifying teeth
* medical disorders requiring prophylactic antibiotic therapy or interfering with the treatment
* periodontal treatment in the past 6 months
* use of drugs known to affect periodontal status (antibiotic, anti-inflammatory, anticonvulsant, immunosuppressant and calcium channel blocker) within the past 6 months
* orthodontic therapy
* pregnancy and lactation
* allergy to metronidazole
* any systemic diseases (e.g.: diabetes and immunological disorders)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in PPD | Change from baseline to 6 months
  Probing pocket depth (PPD) measured from the bottom of the periodontal pocket to the gingival margin were considering four tooth surfaces: mesial, distal, buccal and lingual. Measurements were performed by a calibrated clinician.

SECONDARY OUTCOMES:
Changes in microbiological biofilm composition | Change from baseline to 6 months
  Subgingival biofilm samples were collected from five pockets of each patient, present 5-6mm at the baseline period in a single root tooth.
Changes in VPI | Change from baseline to 6 months
  Visible plaque index (VPI) measured on four tooth surfaces: mesial, distal, buccal and lingual. Measurements were performed by a calibrated clinician.
Changes in GBI | Change from baseline to 6 months
  Gingival bleeding index (GBI) measured on four tooth surfaces: mesial, distal, buccal and lingual. Measurements were performed by a calibrated clinician.
Changes in RAL | Change from baseline to 6 months
  Relative attachment level (RAL) measured from the stent to the bottom of periodontal pocket. Measurements were performed by a calibrated clinician.

OTHER OUTCOMES:
Drug use compliance | After 8 days of periodontal treatment
  Drug use compliance was measured by salivary drug concentration on the eighth day after periodontal debridement.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane C Bergamaschi, PhD, Principal Investigator — University of Campinas, Brazil; Francisco C Groppo, PhD, Study Chair — University of Campinas, Brazil
Locations (1):
- Piracicaba Dental School, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Background] Lorentz TC, Cota LO, Cortelli JR, Vargas AM, Costa FO. Prospective study of complier individuals under periodontal maintenance therapy: analysis of clinical periodontal parameters, risk predictors and the progression of periodontitis. J Clin Periodontol. 2009 Jan;36(1):58-67. doi: 10.1111/j.1600-051X.2008.01342.x. Epub 2008 Oct 30. PMID 19017035
- [Background] Carvalho LH, D'Avila GB, Leao A, Goncalves C, Haffajee AD, Socransky SS, Feres M. Scaling and root planing, systemic metronidazole and professional plaque removal in the treatment of chronic periodontitis in a Brazilian population II--microbiological results. J Clin Periodontol. 2005 Apr;32(4):406-11. doi: 10.1111/j.1600-051X.2005.00720.x. PMID 15811059
- [Background] Moeintaghavi A, Talebi-ardakani MR, Haerian-ardakani A, Zandi H, Taghipour S, Fallahzadeh H, Pakzad A, Fahami N. Adjunctive effects of systemic amoxicillin and metronidazole with scaling and root planing: a randomized, placebo controlled clinical trial. J Contemp Dent Pract. 2007 Jul 1;8(5):51-9. PMID 17618330